CLINICAL TRIAL: NCT03447704
Title: An International, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study of the Efficacy and Safety of BCD-085 (JSC BIOCAD, Russia) in Patients With Active Ankylosing Spondylitis
Brief Title: International Multicenter Comparative Randomized Placebo-controlled Clinical Study of Efficacy and Safety of BCD-085 in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-085-5
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; interleukin 17; monoclonal antibody; netakimab
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — netakimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-085 (netakimab) (Experimental)
  Interventions: Drug: BCD-085
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: BCD-085 — 120 mg of BCD-085 subcutaneously at week 0,1 and 2 every other week
  Other Names: netakimab
  Arms: BCD-085 (netakimab)
Other: placebo — 2 ml of placebo subcutaneously at week 0,1 2 and every other week, starting from week 16 - 120 mg of BCD-085 subcutaneously at week 16,17 and 18 every other week
  Arms: Placebo

SUMMARY:
BCD-085-5 is an International, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study of the Efficacy and Safety of BCD-085. BCD-085 is a monoclonal antibody to interleukin 17. During BCD-085-5 trial patients with active ankylosing spondylitis will receive 120 mg of BCD-085 subcutaneously every other week or placebo up to Week 16. Starting from week 16 all patients will receive BCD-085. Efficacy, PK and safety parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Active ankylosing spondylitis according to modified criteria of New York classification (1984), that was diagnosed at least 3 months prior to screening.
* Active disease according to BASDAI (score 4 or more) if nonsteroidal antiinflammatory drugs were used in the last 3 month prior to screening.
* Mean backache intensity equals 4 points or more.

Exclusion Criteria:

* Total spinal ankylosis.
* Previous treatment with anti-interleukin 17 drugs or anti-interleukin 17 receptor drugs.
* Prior use of >2 biologics to tumor necrosis factor alfa.
* Prior use of live or attenuated vaccines for up to 8 weeks before signing informed consent.
* Prior use of alkylating agents for up to 12 months prior to signing informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
ASAS40 rate at Week 16 | Week 16
  Percentage of patients with ASAS40 response after 16 weeks of therapy (percentage of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40%)

SECONDARY OUTCOMES:
ASAS20 rate | Week 4, 8, 12, 16, 24, 36, 52
  Percentage of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 20%
Change from baseline in BASDAI | Week 4, 8, 12, 16, 24, 36, 52
  Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score in comparison with screening (from 0 to 10). The maximum change is considered to be better outcome
Change from baseline in ASDAS-CRP | Week 4, 8, 12, 16, 24, 36, 52
  Change in ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score Index) score in comparison with screening (from 0 to > 3.5). The maximum change is considered to be better outcome
Change from baseline in SF-36 | Week 16, 36, 52
  Change in SF-36 (The Short Form-36) score in comparison with screening (physical component) (from 15.9 to 62.1). The maximum change is considered to be better outcome
Frequency of AE/SAE | Week 60
  Percentage of patients with AE (adverse events) /SAE (serious adverse events)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JSC BIOCAD
Locations (7):
- Russia (7):
  - Non-governmental Healthcare Institution "Railway Clinical hospital on the Chelyabinsk Station of JSC Russian Railways", Chelyabinsk
  - Chelyabinsk Regional Clinical hospital, Chelyabinsk
  - Kazan State Medical University, Kazan'
  - State Budgetary Higher Vocational Education Institution I.M. Sechenov First Moscow State Medical University, Moscow
  - Omsk Regional Clinical Hospital, Omsk
  - LLC BioEk, Saint Petersburg
  - North-Western State Medical University n.a. I.I.Mechnikov, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mazurov VI, Dubinina TV, Erdes S, Lapshina SA, Soroka NF, Kunder EV, Smirnov AV, Eremeeva AV, Zinkina-Orikhan AV, Morozova MA, Gaydukova IZ. Response to netakimab in radiographic axial spondyloarthritis patients with different baseline C-reactive protein, sacroiliitis evaluated by MRI and peripheral joint involvement status: a post-hoc analysis of the ASTERA study. Clin Exp Rheumatol. 2023 Mar;41(3):718-726. doi: 10.55563/clinexprheumatol/ljpqqe. Epub 2022 Aug 31. PMID 36062743